CLINICAL TRIAL: NCT05754827
Title: Red Blood Cell Distribution Width to Platelet Count Ratio as a Predictor of Cardiovascular Complications in CKD Patients
Brief Title: RDW to Platlet Count Ratio in CKD Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Doha Aly Mohamed, Dr, Sohag University
Other Study IDs: CKD and CV complications
Record Dates: First submitted 2023-02-22; First posted 2023-03-06 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1-CKD patients without cardiovascular complications
  Interventions: Diagnostic Test: RDW to platlet count ratio
- 2-CKD patients with cardiovascular complications
  Interventions: Diagnostic Test: RDW to platlet count ratio

INTERVENTIONS:
Diagnostic Test: RDW to platlet count ratio — RDW to platlet ratio will be measured for all patients and results will be compared between groups

SUMMARY:
The aim of the study is to determine Red blood cell distribution width to platelet count ratio as a predictor of cardiovascular complications in CKD patients

DETAILED DESCRIPTION:
comparative study between RDW to Platlet count ratio in CKD patients without cardiovascular complications and CKD patients with cardiovascular complications

ELIGIBILITY:
* Inclusion Criteria:

  * CKD Patients and patients receive dialysis >18 years old
* Exclusion Criteria:

  * Serious complications of any other organs
  * patients who had previously undergone kidney transplantation .
  * CKD patients with history of previous CVD
  * patients with an infection, blood transfusion or receiving immunosuppressive drugs, as this may have affected the inflammatory response within the 3 months
  * patients who were pregnant
  * patients with chronic hematological disease
  * patient<18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CKD Patients and patients receive dialysis admitted to Sohag University hospital at period of admission 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-04-01 (Estimated); Primary Completion 2024-02-22 (Estimated); Study Completion 2024-03-22 (Estimated)

PRIMARY OUTCOMES:
Comparison of results of RDW to platlet ratio in CKD patients | 1 year
  Calculate RDW to platlet ratio for CKD patints with or without cardiovascular complications and compare the results

REFERENCES:
- [Background] Jankowski J, Floege J, Fliser D, Bohm M, Marx N. Cardiovascular Disease in Chronic Kidney Disease: Pathophysiological Insights and Therapeutic Options. Circulation. 2021 Mar 16;143(11):1157-1172. doi: 10.1161/CIRCULATIONAHA.120.050686. Epub 2021 Mar 15. PMID 33720773